CLINICAL TRIAL: NCT02869334
Title: Remediation of Auditory Recognition in Schizophrenia With Transcranial Direct Current Stimulation (tDCS)
Brief Title: Remediation of Auditory Recognition in Schizophrenia With tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Principal Investigator, Daniel C. Javitt, Professor, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7266
Record Dates: First submitted 2016-07-19; First posted 2016-08-16 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Auditory remediation with active tDCS (Experimental): Auditory remediation program paired with active transcranial direct current stimulation (tDCS) for 30 minutes, 2-3 sessions per week
  Interventions: Device: Active Transcranial direct current stimulation (tDCS); Behavioral: Auditory Remediation
- Auditory remediation with sham tDCS (Experimental): Auditory remediation program paired with sham transcranial direct current stimulation (tDCS) for 30 minutes, 2-3 sessions per week
  Interventions: Device: Sham Transcranial direct current stimulation (tDCS); Behavioral: Auditory Remediation
- Control (computer games with sham tDCS) (Sham Comparator): Non-remediation, control computer activities (e.g. games) with sham transcranial direct current stimulation (tDCS) for 30 minutes, 2-3 sessions per week
  Interventions: Device: Sham Transcranial direct current stimulation (tDCS); Behavioral: Control computer activities

INTERVENTIONS:
Device: Active Transcranial direct current stimulation (tDCS) — Active tDCS, where an extremely weak electric current passes through the brain
  Arms: Auditory remediation with active tDCS
Device: Sham Transcranial direct current stimulation (tDCS) — Sham (inactive or placebo) tDCS
  Arms: Auditory remediation with sham tDCS; Control (computer games with sham tDCS)
Behavioral: Auditory Remediation — Computer program designed to improve discrimination between sounds
  Arms: Auditory remediation with active tDCS; Auditory remediation with sham tDCS
Behavioral: Control computer activities — Computer program (e.g. games), which are not designed to improve discrimination between sounds
  Arms: Control (computer games with sham tDCS)

SUMMARY:
The purpose of this study is to determine whether transcranial direct current stimulation (tDCS), when combined with different forms of computer based training, improves the ability to discriminate small differences between sounds in people diagnosed with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
This study uses an experimental procedure called transcranial direct current stimulation (tDCS). Little is known about how tDCS affects the brain or why some people diagnosed with schizophrenia or schizoaffective disorder have trouble with certain kinds of hearing. This study is being done to see if an experimental computer training program, when combined with tDCS, can help people to hear better. In tDCS, a small amount of electricity is passed through electrodes placed on the head that is able to stimulate the brain. By stimulating the brain, the investigators believe that the functioning of the brain can be altered. This study will test whether such stimulation of the brain, when done with computer training, can improve hearing ability and if this improvement helps in other ways, like detecting changes in someone's tone of voice or understanding other people's emotions better. The data being collected aims to better understand how the brain processes sounds and how tDCS affects the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Primary diagnosis of Schizophrenia or schizoaffective disorder
* English fluency
* Willing/capable to provide informed consent
* Auditory tone matching deficits
* Receiving stable doses of antipsychotic medication(s) for at least 2 weeks
* IQ>75

Exclusion Criteria:

* Serious neurological disorder or medical condition/ treatment known to affect the brain. Neurological Disorder that affects the central nervous system (CNS), such as epilepsy, neurodegenerative disorders, movement disorders and sensory disorders.
* Current or past history (within the last 6 months) of substance abuse or dependence (excluding nicotine)
* Pregnancy or breastfeeding
* Taking anticholinergic medication (e.g. Cogentin, Thorazine, Clozaril, thioridazine)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Javitt, MD, PhD, Principal Investigator — NY State Psychiatric Institute, Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561
- See also: New York State Psychiatric Institute — http://nyspi.org/
- See also: Department of Psychiatry, Columbia University Medical Center — http://columbiapsychiatry.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Auditory Remediation With Active tDCS | Auditory Remediation With Sham tDCS
Started | 10 | 10
Completed | 2 | 3
Not Completed | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auditory Remediation With Active tDCS | Auditory Remediation With Sham tDCS | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (9.9) | 44.7 (14.4) | 42.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5
Tone matching (i.e. ability to match tones following brief delay) [Mean (Standard Deviation); unit: percent correct] | 53.6 (5.1) | 54.3 (12.7) | 54.0 (9.3)

OUTCOME MEASURES:

1. Primary Outcome: Auditory Tone Matching Task
Description: Ability to match tones following brief delay
Time Frame: Change in performance from Baseline at completion of training (week 16)
Population: completers
Measure: Mean (Standard Deviation); unit: %correct, different trials
Arm/Group | Auditory Remediation With Active tDCS | Auditory Remediation With Sham tDCS
Number analyzed (Participants) | 2 | 3
%correct, different trials | -4.3 (12.1) | 4.8 (9.3)

2. Secondary Outcome: Auditory Emotion Recognition (AER) Task
Description: Ability to detect emotion based on tone of voice
Time Frame: Change in performance from Baseline at completion of training (week 16)
Measure: Mean (Standard Deviation); unit: %correct
Arm/Group | Auditory Remediation With Active tDCS | Auditory Remediation With Sham tDCS
Number analyzed (Participants) | 2 | 3
%correct | -3.0 (8.6) | 5.1 (12.2)

3. Secondary Outcome: ER-40
Description: Penn Emotion Recognition Test-40 Faces Version
Time Frame: Change in performance from Baseline at completion of training (week 16)
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Auditory Remediation With Active tDCS | Auditory Remediation With Sham tDCS
Number analyzed (Participants) | 2 | 2
percent correct | -5.0 (3.5) | -1.3 (1.8)

4. Secondary Outcome: The Awareness of Social Inference Test (TASIT)
Description: The TASIT is a measure of social cognition, theory of mind as reflected in the ability to detect lies/sarcasm while viewing social vignettes. Total scores range from 0-100% correct. Higher numbers (positive change) are considered better.
Time Frame: Change in performance from Baseline at completion of training (week 16)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Auditory Remediation With Active tDCS | Auditory Remediation With Sham tDCS
Number analyzed (Participants) | 2 | 3
score on a scale | 10 (4.2) | 0 (6.8)

5. Secondary Outcome: Auditory Mismatch Negativity (MMN)
Description: Change in event related potentials (ERP) acquired during a task of auditory mismatch negativity (MMN), assessed with electroencephalography (EEG)
Time Frame: Change in performance from Baseline at completion of training (week 16)
Population: Subjects who completed post-testing and had usable data
Measure: Mean (Standard Deviation); unit: microvolt
Arm/Group | Auditory Remediation With Active tDCS | Auditory Remediation With Sham tDCS
Number analyzed (Participants) | 1 | 2
microvolt | -1.47 (0) | -.98 (1.07)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Auditory Remediation With Active tDCS | Auditory Remediation With Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/2 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auditory Remediation With Active tDCS (N=2) | Auditory Remediation With Sham tDCS (N=3)
sedation (Nervous system disorders) | 1 (1) | 0 (0) — Moderate sedation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT02869334/Prot_SAP_000.pdf